CLINICAL TRIAL: NCT01689961
Title: Be Healthy in Pregnancy (BHIP) With Nutrition and Exercise
Acronym: BHIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Agriculture and Agri-Food Canada (Other Government); Dairy Farmers of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 12-469
Record Dates: First submitted 2012-09-13; First posted 2012-09-21 (Estimated); Last update posted 2020-10-01 (Actual); Status verified 2019-03

CONDITIONS: Pregnancy Complications; Weight Gain
Keywords: Nutrition; Physical activity; Gestational weight gain; Pregnancy outcomes; Birth
MeSH Terms: conditions — Pregnancy Complications; Weight Gain; Motor Activity; Gestational Weight Gain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutrition+Exercise Intervention (Experimental): Structured + monitored nutrition and exercise intervention:
  The exercise intervention includes a custom-designed pregnancy-specific group walking class of 30-60 min. 1x/week and a prescribed at-home walking program for 10,000 steps/day. The nutrition intervention is a high protein (25% energy) low-fat dairy food plan designed to meet energy needs and with individualized counselling. The intervention will include 2 x/month weight monitoring and records of nutrition and activity to ensure adherence
  Interventions: Behavioral: Structured + monitored nutrition and exercise intervention
- Usual Prenatal Care (No Intervention): Mothers in the Control Group will be followed by their primary care provider and have usual access to public health services. In addition, they will be asked to attend 2 focus group sessions exploring women's experiences with exercise, nutrition, and weight gain in pregnancy. Women will receive information about healthy pregnancy from Health Canada.

INTERVENTIONS:
Behavioral: Structured + monitored nutrition and exercise intervention — The exercise intervention includes a custom-designed pregnancy-specific group walking class of 30-60 min. 1x/week and a prescribed at-home walking program for 10,000 steps/day. The nutrition intervention is a high protein (25% energy) low-fat dairy food plan designed to meet energy needs and with individualized counselling. The intervention will include 2 x/month weight monitoring and records of nutrition and activity to ensure adherence.
  Arms: Nutrition+Exercise Intervention

SUMMARY:
Excess weight gain in pregnancy is a major problem affecting 55-75% of Canadian women who enter pregnancy overweight or obese and about 40% of women who are normal weight. Excess weight gain puts mothers at risk for health problems such as diabetes and developing or sustaining obesity after pregnancy, and puts their babies at risk of being born too large or developing related health problems. Mothers will be randomized to a structured high dairy protein diet and walking program or the usual care by their care provider. The investigators research questions are: Will a structured nutrition and exercise program in pregnancy compared to usual prenatal care increase the chance that mothers will achieve pregnancy weight gain within the current recommendations; improve health measures, in mother and infant at six months post-partum; to evaluate the benefits of a high dairy intake in pregnancy on maintenance of bone status in the mother and bone health outcomes in the child in early life (6 months); and to investigate the interactions between genes associated with bone health and high dairy diet supplementation on bone status in mothers during pregnancy, and bone health in mothers post-delivery and children to 6 months of age. Mothers' weight, physical activity and adherence to the nutrition plan will be assessed until birth and at follow-up with their infants at 6 months after birth. The research team will ensure new information is quickly transferred to programs to assist women to have healthier pregnancies.

DETAILED DESCRIPTION:
This will be a 2-arm randomized 3-site trial. Recruitment will be within the community care clinics by poster and flyer advertisements. Pregnant women will be stratified by BMI categories and study site and randomized within strata to Group A (Nutrition+Exercise intervention program) or Group B (Usual Prenatal Care + Health Canada materials about healthy pregnancy + two focus group sessions exploring women's experiences with exercise, nutrition and weight gain in pregnancy).

Primary research question: Among pregnant women, does introducing a structured and monitored nutrition and exercise program (treatment) in early pregnancy compared with Usual Prenatal Care (control) increase the likelihood of attaining gestational weight gain within the Institute of Medicine (IOM) guidelines over the pregnancy period? Secondary research questions: Among pregnant women (population), does introducing a structured and monitored nutrition and exercise program in early pregnancy (intervention) compared with Standard Prenatal Care (control) lead to 1) better maternal outcomes (outcome) at 6 months post- partum; and ii) better infant outcomes (outcome) at 6 months post partum?; and 2) i) to evaluate the benefits of a high dairy intake in pregnancy on maintenance of bone status in the mother and bone health outcomes in the child in early life (6 months); and ii) to investigate the interactions between genes associated with bone health and high dairy diet supplementation on bone status in mothers during pregnancy, and bone health in mothers post-delivery and children to 6 months of age.

Experimental and Control groups: Both groups of mothers and their health care providers will be given the Health Canada materials on "Healthy Weight Gain during Pregnancy", "Eating Well with Canada's Food Guide" and the "Pregnancy Weight Gain Calculator". Baseline information will be recorded for eligible and consenting women after which they will be randomized to Experimental or Control group. Nutrition intake, physical measures and physical activity will be recorded at baseline, 26-28 weeks, 36-38 weeks of gestation, and 6 months postpartum in the same manner for both groups. All mothers will receive the study promotional materials and small incentives. Also, all mothers will be followed by their primary care provider and have usual access to public health.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant females > 18 years of age with singleton pregnancies (either nulliparous or multiparous);
* less than 17 weeks gestation;
* a pre pregnancy BMI < 40 kg/m2 (owing to the fact that severe obesity with BMI> 40 may have limitations with respect to physical activity);
* plans to deliver at a Hamilton or London regional hospital or by home birth and willing to attend research visits at the community site where they were recruited;
* able to tolerate dairy foods;
* approval of primary care provider;
* able to provide signed informed consent.

Exclusion Criteria:

* unable to understand some English;
* type 1 or type 2 diabetes;
* known contraindications to exercise as recommended by the Canadian clinical practice guidelines for pregnancy;
* severe gastrointestinal diseases or conditions;
* any significant heart, kidney, liver or pancreatic diseases;
* pre-existing diabetes;
* currently smoking;
* a depression score 12 or above on the validated Edinburgh depression questionnaire.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 242 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Gestational weight gain within IOM guidelines | Change from baseline at 38 weeks gestation
  Among pregnant women (population), does introducing a structured and monitored nutrition and exercise program (treatment) in early pregnancy compared with Usual Prenatal Care (control) increase the likelihood of attaining gestational weight gain within the IOM guidelines (outcome) over the pregnancy period?

SECONDARY OUTCOMES:
Maternal and infant outcomes | 6 months postpartum
  The secondary research question is whether the proposed intervention will result in i) better maternal outcomes (outcome) at 6 months post- partum; and ii) better infant outcomes (outcome) at 6 months post partum?
Bone health of mother and baby | 6 months post-partum
  In mother: plasma/serum measures of bone mineralization and bone resorption and vitamin D status; bone mineral density as measured by dual energy x-ray absorptiometry scan.
  In infant: bone mineral content as measured by dual energy x-ray absorptiometry scan.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie A Atkinson, PhD, Principal Investigator — McMaster University
Locations (4):
- Canada (4):
  - Burlington Midwives Clinic, Burlington, Ontario
  - McMaster Family Health Team, Hamilton, Ontario
  - Hamilton Midwives Clinics, Hamilton, Ontario
  - Exercise and Pregnancy Laboratory, London, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krzeczkowski JE, Mortaji N, Atkinson S, Schmidt LA, Van Lieshout RJ. Adaptive changes in multiple aspects of emotion regulation in the offspring of pregnant persons receiving a diet-and-exercise intervention relative to usual pregnancy care: a randomized controlled trial. Am J Clin Nutr. 2025 Jan;121(1):50-59. doi: 10.1016/j.ajcnut.2024.10.022. Epub 2024 Oct 30. PMID 39486684
- [Derived] Mortaji N, Krzeczkowski J, Atkinson S, Amani B, Schmidt LA, Van Lieshout RJ. Early neurodevelopment in the offspring of women enrolled in a randomized controlled trial assessing the effectiveness of a nutrition + exercise intervention on the cognitive development of 12-month-olds. J Dev Orig Health Dis. 2023 Aug;14(4):532-539. doi: 10.1017/S204017442300020X. Epub 2023 Jul 14. PMID 37448202
- [Derived] Dempsey K, Mottola MF, Atkinson SA. Comparative Assessment of Diet Quality and Adherence to a Structured Nutrition and Exercise Intervention Compared with Usual Care in Pregnancy in a Randomized Trial. Curr Dev Nutr. 2023 May 13;7(6):100097. doi: 10.1016/j.cdnut.2023.100097. eCollection 2023 Jun. PMID 37441683
- [Derived] Mortaji N, Krzeczkowski J, Atkinson S, Amani B, Schmidt LA, Van Lieshout R. Preliminary findings of emotion regulation in 12-month-old infants of mothers enrolled in a randomized controlled trial assessing a nutrition + exercise intervention. Dev Psychobiol. 2023 Mar;65(2):e22376. doi: 10.1002/dev.22376. PMID 36811372
- [Derived] Shanmuganathan M, Bogert M, Kroezen Z, Britz-McKibbin P, Atkinson SA. Dynamic Metabolic Signatures of Choline and Carnitine across Healthy Pregnancy and in Cord Blood: Association with Maternal Dietary Protein. J Nutr. 2023 Apr;153(4):999-1007. doi: 10.1016/j.tjnut.2023.02.013. Epub 2023 Feb 11. PMID 36780943
- [Derived] Perreault M, Mottola MF, Atkinson SA; BHIP study team. Individualized high dairy protein + walking program supports bone health in pregnancy: a randomized controlled trial. Am J Clin Nutr. 2022 Oct 6;116(4):887-896. doi: 10.1093/ajcn/nqac182. PMID 35759368
- [Derived] Murray-Davis B, Grenier L, Atkinson SA, Mottola MF, Wahoush O, Thabane L, Xie F, Vickers-Manzin J, Moore C, Hutton EK. Experiences regarding nutrition and exercise among women during early postpartum: a qualitative grounded theory study. BMC Pregnancy Childbirth. 2019 Oct 21;19(1):368. doi: 10.1186/s12884-019-2508-z. PMID 31638920
- [Derived] Perreault M, Atkinson SA, Mottola MF, Phillips SM, Bracken K, Hutton EK, Xie F, Meyre D, Morassut RE, Prapavessis H, Thabane L; BHIP Study team. Structured diet and exercise guidance in pregnancy to improve health in women and their offspring: study protocol for the Be Healthy in Pregnancy (BHIP) randomized controlled trial. Trials. 2018 Dec 19;19(1):691. doi: 10.1186/s13063-018-3065-x. PMID 30567604